CLINICAL TRIAL: NCT01529008
Title: Phase 3, Pivotal, Multicentre, Randomised, Double-blind Controlled Study to Evaluate the Efficacy and Safety of Autologous Osteoblastic Cells (PREOB®) Implantation in Early Stage Non Traumatic Osteonecrosis of the Femoral Head
Brief Title: Study on Autologous Osteoblastic Cells Implantation to Early Stage Osteonecrosis of the Femoral Head
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: the interim results suggest that it is unlikely that the primary objective will be achieved at the final analysis
Sponsor: Bone Therapeutics S.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PREOB-ON3
Record Dates: First submitted 2012-02-02; First posted 2012-02-08 (Estimated); Results first posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Osteonecrosis of the Femoral Head
Keywords: Osteonecrosis; Femoral Head; Hip; Orthopedics; Bone; Musculoskeletal Disorders
MeSH Terms: conditions — Legg-Calve-Perthes Disease; Osteonecrosis; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Core decompression/PREOB® implantation (Experimental)
  Interventions: Drug: Core decompression/PREOB® implantation
- Core decompression/placebo implantation (Placebo Comparator)
  Interventions: Drug: Core decompression/placebo implantation

INTERVENTIONS:
Drug: Core decompression/PREOB® implantation — All patients will undergo a core decompression under general anesthesia combined with the implantation of PREOB® into the necrotic lesion (single administration).
  Arms: Core decompression/PREOB® implantation
Drug: Core decompression/placebo implantation — All patients will undergo a core decompression under general anesthesia combined with the implantation of placebo into the necrotic lesion (single administration).
  Arms: Core decompression/placebo implantation

SUMMARY:
Non-traumatic osteonecrosis is a painful disorder of the hip characterized by a necrosis of the osteomedullary tissue, which leads to subchondral bone collapse and joint destruction. Core decompression is currently the treatment of choice for early stage osteonecrosis of the femoral head. This method consists in decompressing the rigid intra-osseous chamber to promote revascularization, thus halting progression of the disease and stimulating repair. Still this treatment remains highly controversial, since the success rates of the first studies have not been repeated.

The exact pathology mechanisms involved in osteonecrosis have not yet be fully elucidated. Several hypotheses have been evoked, including fat embolism, trabecular bone microfractures, microvascular tamponade and, more recently, impaired bone and/or mesenchymal cells recruitment.

Three studies have indicated the potential clinical benefits of cell-based approaches for the treatment of osteonecrosis (Hernigou 1997, Hernigou & Beaujean 2002, Gangji et al. 2004). This is on the basis of these observations that a proprietary population of autologous osteoblastic cells (PREOB®) has been developed.

This Phase 3 study aims at demonstrating the efficacy and safety of PREOB® in the treatment of early stage osteonecrosis of the femoral head. More specifically, the purpose of the study is to demonstrate that core decompression/PREOB® implantation into the necrotic lesion is superior to core decompression/placebo implantation in relieving hip symptoms and halting (or reverting) radiological progression of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between 18 and 70 years (inclusive) with a diagnosis of ARCO Stage I or II non-traumatic osteonecrosis of the femoral head, confirmed by central imaging analysis based on X-ray and MRI.
* Ability to provide a written, dated, and signed informed consent prior to any study related procedure and to understand and comply with study requirements
* Diagnosis of Osteonecrosis:

  1. ARCO stage I associated with WOMAC® VA3.1 pain score ≥20 mm and necrotic angle sum ≥190° based on sagittal and coronal MRI views or
  2. ARCO stage II associated with WOMAC® VA3.1 pain score ≥20 mm if necrotic angle sum <190° based on sagittal and coronal MRI views or
  3. ARCO stage II associated or not with pain if necrotic angle sum is ≥190° based on sagittal and coronal MRI views
  4. Associated with corticosteroid and/or with alcohol abuse and/or idiopathic
* Normal haematology function, defined as leukocytes ≥3000/mm3, absolute neutrophils count ≥1500/mm3, platelets ≥140,000/mm3, and haemoglobin concentration ≥10g/dl (peripheral blood test)

Exclusion Criteria:

Current symptoms and/or signs related to the disease under study

* Exclusively diaphyseal or metaphyseal osteonecrotic lesion
* Traumatic or hyperbaric osteonecrosis, or osteonecrosis associated with hemoglobinopathy or coagulopathy (e.g., thalassemia, sickle cell disease,…), or Gaucher's disease
* Any other focal or diffuse bone marrow lesion
* Osteoarthritis at the target hip defined as Kellgrens stage ≥2, as assessed by the Central Radiologist
* Patients suffering from any medical conditions interfering with patient's pain evaluation of the hip under evaluation, such as knee arthritis.
* Bone fracture or bone infection at hip under evaluation.
* Patients who are candidates for any predictable joint replacement on the hip that is evaluated Current or previous diagnoses, signs and/or symptoms
* Active hepatitis B (defined as positive HBs Ag and/or positive PCR), or active hepatitis C (defined as positive PCR), positive serology for HIV, or Syphilis, or HTLV-1, and any other tests that may be required by the authorities in case of a new disease outbreak that can affect the safety of the physicians and operators at the time of patient screening.
* Presence, or previous history, of risks factors for diseases caused by prions, and recipients of grafts of cornea, sclera, and dura mater
* History of blood loss exceeding 450 ml (incl. donations) within 1 month of screening
* Renal impairment defined by an estimated creatinine clearance value < 30 ml per min, calculated with the Cockcroft-Gault formula
* Hepatic impairment, defined as alanine aminotransferase or aspartate aminotransferase ≥ 3 times the upper limit of normal
* Poorly controlled diabetes mellitus, defined as HbA1C > 9%
* Global sepsis
* Allergy to gentamicin or porcine collagen or any substance or device the patient might be exposed to in the context of the study related interventions (i.e., bone marrow harvesting and implantation), as judged by the Investigator
* History of hypersensitivity to human biological material, including blood and blood derived products, documented clinically or by laboratory tests
* Current or past history of solid or haematological neoplasia (except for basal cell carcinoma of the skin and for carcinoma in situ of the cervix that has been treated with no evidence of recurrence)
* History of bone marrow transplantation
* Patients with a life expectancy less than 2 years, as judged by the Investigator Current or previous treatment
* Patients having participated in another clinical trial within 3 months of screening
* Patients previously treated with PREOB®
* Patients treated by core decompression of the hip under evaluation within 6 months of screening
* Treatment with doses of prednisolone ≥15 mg per day (or equivalent) within 1 month from screening, and patients with anticipated needs of daily corticoid doses ≥15 mg prednisone (or equivalent) in the 6 -month period following PREOB/Placebo implantation
* Illicit drug or alcohol abuse interfering with patient's ability to understand and comply with study requirements, as judged by the Investigator

Safety aspects concerning female patients of childbearing potential

* Pregnancy
* Breast-feeding
* Women with childbearing potential not willing or able to use reliable contraceptive method for at least 6 weeks prior to screening and during the whole study period. Reliable contraceptive methods include orally administered hormonal contraceptives, surgical intervention (e.g., tubal ligation), and intrauterine device (IUD).

Other exclusion criteria:

* Body Mass Index (BMI) ≥ 35 kg/m2
* Patients unable to undergo MRI, e.g. patients with pace-maker, intra-ocular or intra-cerebral metallic foreign bodies, and mechanical artificial heart valves
* Patients unable to undergo general anaesthesia or surgical intervention

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-11; Primary Completion 2017-05 (Actual); Study Completion 2018-11 (Actual)

REFERENCES:
- [Derived] Jayankura M, Thomas T, Seefried L, Dubrana F, Gunther KP, Rondia J, Davis ET, Winnock de Grave P, Carron P, Gangji V, Vande Berg B, Godeaux O, Sonnet W. Does Adjunction of Autologous Osteoblastic Cells Improve the Results of Core Decompression in Early-stage Femoral Head Osteonecrosis? A Double-blind, Randomized Trial. Clin Orthop Relat Res. 2023 Aug 1;481(8):1527-1540. doi: 10.1097/CORR.0000000000002610. Epub 2023 Mar 24. PMID 36961220

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: the Data Safety Monitoring Board recommended that the study be stopped for futility
Period: Screening
Arm/Group | Core Decompression/PREOB® Implantation | Core Decompression/Placebo Implantation
Started | 35 | 33
Completed | 35 | 33
Not Completed | 0 | 0
Period: Bone Marrow Harvesting
Arm/Group | Core Decompression/PREOB® Implantation | Core Decompression/Placebo Implantation
Started | 35 | 33
Completed | 34 | 30
Not Completed | 1 | 3
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2
Period: Treatment
Arm/Group | Core Decompression/PREOB® Implantation | Core Decompression/Placebo Implantation
Started | 34 | 30
Completed | 25 | 29
Not Completed | 9 | 1
Not completed — Adverse Event | 6 | 0
Not completed — Other | 3 | 1
Period: Efficacy Analysis
Arm/Group | Core Decompression/PREOB® Implantation | Core Decompression/Placebo Implantation
Started | 25 | 29
Completed | 23 | 26
Not Completed | 2 | 3
Not completed — Protocol Violation | 2 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Core Decompression/PREOB® Implantation | Core Decompression/Placebo Implantation | Total
Number analyzed (Participants) | 34 | 30 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (9.9) | 45.4 (9.7) | 45.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 27 | 26 | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnic origin: Caucasian/White | 30 | 29 | 59
  Ethnic origin: Black | 2 | 1 | 3
  Ethnic origin: Oriental/Asian | 1 | 0 | 1
  Ethnic origin: Hispanic | 0 | 0 | 0
  Ethnic origin: Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Treatment Responders
Description: A patient was considered as having responded to treatment if:
  * the WOMAC VA3.1 pain subscale score (Western Ontario and McMaster Universitie Visual Analogue scale) of the study treated hip improved from baseline by at leat the MCID (minimal clinically important difference ) the WOMAC VA3.1 pain subscale score is Visual score based on 10 cm and
  * the study treated hip did not progress to fractural stages (ARCO III or higher) as assessed by conventional X-ray
Time Frame: 24 months
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of treatment responders
Arm/Group | Core Decompression/PREOB® Implantation | Core Decompression/Placebo Implantation
Number analyzed (Participants) | 23 | 26
percentage of treatment responders | 60.9 [38.5 to 80.3] | 69.2 [48.2 to 85.7]
Statistical Analysis 1: Comparison: Core Decompression/PREOB® Implantation vs Core Decompression/Placebo Implantation; Test type: Superiority; p = 0.539, Fisher Exact; Proportion treatment responder Differenc = -0.08, 95% CI 2-sided [-0.35 to 0.18] — Percentage of treatment responders in PREOB® group is 60.9% ((14/23)*100), compared with 69.2% ((18/26)*100) in Placebo. Difference in percentage is -8.3 Difference in treatment responders proportion: PREOB® (0.609) - Placebo (0.692) = -0.08

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Core Decompression/PREOB® Implantation | Core Decompression/Placebo Implantation
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/29
Serious Adverse Events (participants affected / at risk) | 16/25 | 18/29
Other Adverse Events (participants affected / at risk) | 22/25 | 25/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Decompression/PREOB® Implantation (N=25) | Core Decompression/Placebo Implantation (N=29)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
disease progression (General disorders) | 7 (9) | 14 (17)
Chest pain (General disorders) | 1 (1) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 2 (2) | 0 (0)
non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Breathing-related sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Apendicitis (Infections and infestations) | 1 (1) | 0 (0)
Campylobacter Infection (Infections and infestations) | 1 (1) | 0 (0)
Cholangitis Infective (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Acute renal kidney (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Hip Arthroplasty (Social circumstances) | 1 (1) | 0 (0)
Removal of internal fixation (Surgical and medical procedures) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (2)
Bile duct stenosis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Lung transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
Transplant evaluation (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angiodema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Decompression/PREOB® Implantation (N=25) | Core Decompression/Placebo Implantation (N=29)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (18) | 13 (19)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Pain (General disorders) | 1 (1) | 2 (2)
Systemic Inflammatory Response Syndrome (General disorders) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 4 (4) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT01529008/Prot_SAP_000.pdf